CLINICAL TRIAL: NCT05972681
Title: A Randomized Controlled Trial of Bupivacaine With Epinephrine for Local Pain Control Following Perineal Laceration Repair in Patients With Pre-existing Epidural Analgesia: The PAIN Trial
Brief Title: The PAIN (Pelvic Area Injection for Numbness) Study
Acronym: PAIN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-14825
Record Dates: First submitted 2023-07-17; First posted 2023-08-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Vaginal Laceration During Delivery
MeSH Terms: interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be blinded to the patient, the nurse carrying for the patient and providing the randomized, unlabeled syringe, the provider performing the perineal repair, the research team asking the maternal satisfaction questions, and the researcher analyzing the data. To assure blinding, the selection of the medication given, and the preparation of such medication will be performed by the labor and delivery anesthesia team. No one involved directly in the perineal laceration repair, or obtaining research information, nor the patient, will know what was injected. Subject treatment assignments will remain blinded until the final subject has completed follow up and all data has been recorded and validated. Urgent, immediate unblinding due to medical emergency may be authorized by the Investigator. When possible, the treatment assignment will be provided to the treating physician to maintain the blind for the Investigator and study staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Local Anesthesia arm (Experimental): Bupivicaine and Epinephrine
  Interventions: Drug: Bupivacaine; Drug: Epinephrine
- Normal saline sham arm (Sham Comparator)
  Interventions: Other: Sham normal saline arm

INTERVENTIONS:
Drug: Bupivacaine — 10 milliliters (ml) of bupivacaine 0.50% injected to the vaginal laceration site.
  Arms: Local Anesthesia arm
Drug: Epinephrine — Epinephrine (1:200,000) injected to the vaginal laceration site.
  Arms: Local Anesthesia arm
Other: Sham normal saline arm — 10 milliliter (ml) of normal saline injected to the vaginal laceration site.
  Arms: Normal saline sham arm

SUMMARY:
Postpartum pain can interfere with patient's ability to care for themselves, and their newborn, and untreated pain is associated with risk of greater opioid use, postpartum depression, and development of persistent pain. The research hypothesis of this study is that adding a locally injected analgesic, which will take effect once the epidural analgesia fades, may alleviate perineal pain and improve women's overall well-being and satisfaction.

The objective of this study is to determine if prolonged analgesia and higher rate of maternal satisfaction are found when bupivacaine with epinephrine infiltration is used for perineal repair as compared to sham injection in patients with pre-existing effective epidural analgesia at time of perineal laceration repair.

DETAILED DESCRIPTION:
Perineal lacerations, the disruption of the skin, mucosa and sometimes muscles that happen commonly during vaginal birth secondary to stretching of the introitus; are present in more than 75% of all vaginal deliveries. These lacerations can be classified based on the location and depth (layers injured). However, the classification of these lacerations does not correlate necessarily with postpartum pain. Severe lacerations, as those compromising the external or internal anal sphincter are less common and associated with more postpartum pain.

It is common practice that only those lacerations causing bleeding, or distortion of normal pelvic anatomy are repaired. The repair of such lacerations at Montefiore Einstein is usually done using lidocaine for non-epiduralized patients; however, for patients with a functional epidural, no anesthetic agents are given locally to aid on long term pain control.

The prevalence of perineal lacerations is more than 75% of all vaginal deliveries. The repair of such lacerations in the institution is usually done using lidocaine for non-epiduralized patients versus no local injection in patients with a pre-existing epidural analgesia. The prevalence of epidural analgesia use among women who underwent vaginal delivery in cross-sectional study of over 2 million deliveries in the United States was 71.1%. Once the analgesic effect of the epidural analgesia fades, the laceration may cause uncontrolled postpartum pain which can affect both the physical and mental recovery period, extend hospital stays, and increase the potential for serious adverse reactions with pain medications.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* Healthy with a singleton pregnancy
* English or Spanish speaking
* Ongoing functioning epidural throughout the laceration repair
* Multiparous or nulliparous
* Ability to consent for themselves

Exclusion Criteria:

* Underwent an operative vaginal delivery and whose vaginal delivery was complicated by a postpartum hemorrhage
* Vaginal delivery was complicated by a postpartum hemorrhage
* Have multiple gestations
* Complaints of non-functional epidural
* Allergic to bupivacaine and/or epinephrine
* Epidural was a combined spinal-epidural (CSE)
* Received an epidural top-off (bolus of local anesthetic injected into the epidural catheter) < 3 hours from the perineal repair
* Experienced extreme pain at time of study consent (pain scale score > 3 on 0-10 scale)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesic | Up to 24 hours after perineal laceration
  Average time to first analgesic (TFA) will be evaluated per patient as the duration interval following injection to administration of the first analgesic, as applicable.
Maternal Satisfaction | 24 hours after perineal laceration
  Maternal satisfaction will be assessed by participants' rating their ability to carry out their daily living activities at 24hrs using a 4-point scale (very poor; poor; good; or very good)
Maternal Satisfaction | 48 hours after perineal laceration
  Maternal satisfaction will be assessed by participants' rating their ability to carry out their daily living activities at 24hrs using a 4-point scale (very poor; poor; good; or very good)
Maternal Satisfaction | 7 days after perineal laceration
  Maternal satisfaction will be assessed by participants' rating their ability to carry out their daily living activities at 24hrs using a 4-point scale (very poor; poor; good; or very good)
Pain score after injection at perineal laceration | Immediately and 24 hours after perineal laceration
  Participants will self-report measures of symptoms using the Visual Analog Scale (VAS) to determine acute and chronic pain. Participants record a single handwritten mark at one point along the length of a 10-cm line that represents a continuum between the two ends of a scale where "no pain" is on the left end (0 cm) of the scale and the "worst pain" is on the right end of the scale (10 cm). Measurements from the starting point (left end) of the scale to the patients' marks are recorded in centimeters and are interpreted as the intensity of pain. The values will be used to track pain progression for a patient and to compare pain between patients with similar conditions

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Estrada, MD, FACOG, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goh R, Goh D, Ellepola H. Perineal tears - A review. Aust J Gen Pract. 2018 Jan-Feb;47(1-2):35-38. doi: 10.31128/AFP-09-17-4333. PMID 29429318
- [Background] Butwick AJ, Bentley J, Wong CA, Snowden JM, Sun E, Guo N. United States State-Level Variation in the Use of Neuraxial Analgesia During Labor for Pregnant Women. JAMA Netw Open. 2018 Dec 7;1(8):e186567. doi: 10.1001/jamanetworkopen.2018.6567. PMID 30646335
- [Background] Dengler KL, Simpson KJ, Strauchon CJ, Shaddeau AK, Brooks DI, Gruber DD. A randomized controlled trial of liposomal bupivacaine for pain following obstetrical laceration. Am J Obstet Gynecol MFM. 2020 Aug;2(3):100115. doi: 10.1016/j.ajogmf.2020.100115. Epub 2020 Apr 15. PMID 33345866
- [Background] Pharmacologic Stepwise Multimodal Approach for Postpartum Pain Management: ACOG Clinical Consensus No. 1. Obstet Gynecol. 2021 Sep 1;138(3):507-517. doi: 10.1097/AOG.0000000000004517. PMID 34412076
- [Background] Schinkel N, Colbus L, Soltner C, Parot-Schinkel E, Naar L, Fournie A, Granry JC, Beydon L. Perineal infiltration with lidocaine 1%, ropivacaine 0.75%, or placebo for episiotomy repair in parturients who received epidural labor analgesia: a double-blind randomized study. Int J Obstet Anesth. 2010 Jul;19(3):293-7. doi: 10.1016/j.ijoa.2009.11.005. Epub 2010 Jun 2. PMID 20627696
- [Background] Deshpande JP, Saundattikar GY. Lignocaine Versus Ropivacaine Infiltration for Postpartum Perineal Pain. Anesth Essays Res. 2017 Apr-Jun;11(2):300-303. doi: 10.4103/0259-1162.177191. PMID 28663610
- [Background] Mahajan A, Derian A. Local Anesthetic Toxicity. StaPearls. Bookshelf ID: NBK499964. PMID: 29763139